CLINICAL TRIAL: NCT00588796
Title: Alteration in Fibrinogen Metabolism in Patients With Severe Burns and Traumatic Injuries
Brief Title: Study of Fibrinogen Metabolism During Severe Trauma and Burns
Status: Completed | Type: Observational
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: H-04-017
Record Dates: First submitted 2007-12-25; First posted 2008-01-09 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Burn Injury; Major Trauma
Keywords: fibrinogen; burns; trauma; metabolism
MeSH Terms: conditions — Burns; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy Volunteers: Healthy Volunteers
- Burn patients: Patients who have sustained burn injury greater than or equal to 20% of total body surface area
- Trauma patients: Patients who have undergone trauma

SUMMARY:
To study the fibrinogen metabolic changes in relation to coagulation disorder in patients with severe burns and trauma injuries. As a result of the burn or trauma injury breakdown of fibrinogen is accelerated.

DETAILED DESCRIPTION:
In this protocol, we will investigate fibrinogen metabolism in burn and trauma patients, using an 8h infusion of stable isotopes labeled amino acids (1-13C-phenylalanine, 2H5-phenylalanine, and 2H3-ketoisocaporate). The increase of the labeled amino acids incorporating into fibrinogen during the infusion and the decay of labeled fibrinogen after stopping the isotopes infusion (as measured by GC-MS) will be used to calculate fibrinogen synthesis and degradation. Stable isotopes are non-radioactive.

ELIGIBILITY:
Inclusion Criteria:

* 20% total body surface area burn or more
* severe trauma with injury severity score greater than 10
* between ages of 18 and 65 years

Exclusion Criteria:

* history of blood clotting disorder
* history of liver disease such as cirrhosis or hepatitis
* pregnant or nursing
* allergic to iodine, shellfish or dye used in X-Rays
* taking long term medications for blood clotting usch as Coumadin or Plavix
* prisoners
* receiving total parenteral nutrition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Burn patients Trauma patients Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2005-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
During the flow phase following burn or trauma injury, fibrinogen degradation is accelerated | 7

SECONDARY OUTCOMES:
Fibrinogen degradation stimulates fibrinogen synthesis at the expense of whole body protein catabolism | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Wenjun Z Martini, PhD, Principal Investigator — United States Army Institute of Surgical Research

REFERENCES:
- [Background] Zuckerman L, Caprini JA, Lipp V, Vagher JP. Disseminated intravascular multiple systems activation (DIMSA) following thermal injury. J Trauma. 1978 Jun;18(6):432-9. doi: 10.1097/00005373-197806000-00008. PMID 660699